CLINICAL TRIAL: NCT00932932
Title: 11 Beta Hydroxysteroid Dehydrogenase 1 (11-beta HSD 1) Activity in Patients With Prader-Willi Syndrome and in Healthy Controls
Brief Title: Cortisol Activity in Patients With Prader-Willi Syndrome and Healthy Controls
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Jill Jacobson,MD, Children's Mercy Hospitals and Clinics
Other Study IDs: 09 01-014
Record Dates: First submitted 2009-07-02; First posted 2009-07-07 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Prader-Willi Syndrome
MeSH Terms: conditions — Prader-Willi Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- PWS not receiving Growth Hormone
- Control subjects healthy or obese
- PWS subjects starting Growth Hormone

SUMMARY:
The purpose of the study is to find out if people with Prader-Willi syndrome have a difference in the protein which changes inactive cortisone to the active stress hormone cortisol.

ELIGIBILITY:
Inclusion Criteria:

* Prader-Willi syndrome confirmed by molecular testing, ages 6 months to adult
* Controls: Age-matched, sex-matched, developmentally normal, BMI-controlled healthy or obese subjects

Exclusion Criteria:

* PWS subjects without molecular confirmation of the diagnosis
* Subjects receiving glucocorticoid treatment within 3 months of evaluation
* Subjects receiving growth hormone within one year prior to analysis

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Defined population
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2009-02; Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Moore, MD, Principal Investigator — Children's Mercy Hospital Kansas City